CLINICAL TRIAL: NCT05017376
Title: Evaluating the Effect of Optical Zones on Myopia and Astigmatism Correction in SMILE: Vector Analysis
Brief Title: Evaluating the Effect of Optical Zones on Correction for SMILE: Vector Analysis
Status: Completed | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TJYYLL-202034
Record Dates: First submitted 2021-08-11; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Myopia
Keywords: small incision lenticule extraction; vector analysis
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: small optical zone
  Interventions: Procedure: small incision lenticular extraction
- group B: large optical zone
  Interventions: Procedure: small incision lenticular extraction

INTERVENTIONS:
Procedure: small incision lenticular extraction — In patients with the same degree of myopia, different optical zones were designed for operation

SUMMARY:
Evaluate the effect of the size of optical zones (OZ) on myopia and astigmatism correction in small incision lenticular extraction.

DETAILED DESCRIPTION:
To retrospectively study whether different surgical optical zone sizes affect the correction of diopter and astigmatism in myopia patients. Divided into 2 groups according to the diameter of the optical zone. The vector analysis method was used to analyze the changes and errors of astigmatism in TR and SIR after operation. Generalized Estimation Equation (GEE) model is used for multiple regression analysis to evaluate the potential factors related to the error value.

ELIGIBILITY:
Inclusion Criteria:

* no ocular conditions
* normal topography
* central corneal thickness, >500µm
* residual stromal thickness, >280 µm
* pupil diameter, 2.78-4.9 mm (average, 3.76±0.43 mm);

Exclusion Criteria:

* history of intraocular surgery
* pupil diameter, >4.9 mm or <2.78mm
* keratoconus or corneal ectasia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: age of patients between 18-45 years; spherical refraction of -3.00 to -6.00 diopters (D) with or without astigmatism (<-3.00 D); spherical equivalent, -3.00 to -6.00 D; corrected distant visual acuity (CDVA), >20/25
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
astigmatic changes | 2021.03
  Observe the effect on changes in astigmatism by target induced astigmatism (TIA) versus surgically induced astigmatism (SIA)
error value | 2021.04
  Target refraction (TR) and surgically induced refraction (SIR) under different optical zones

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, Study Chair — Tianjin Eye Hospital
Locations (1):
- Tianjin Eye Hospital, Tianjin, China

REFERENCES:
- [Result] Moshirfar M, Thomson AC, West WB Jr, Hall MN, McCabe SE, Thomson RJ, Ronquillo YC, Hoopes PC. Initial Single-Site Experience Using SMILE for the Treatment of Astigmatism in Myopic Eyes and Comparison of Astigmatic Outcomes with Existing Literature. Clin Ophthalmol. 2020 Oct 29;14:3551-3562. doi: 10.2147/OPTH.S276899. eCollection 2020. PMID 33154614
- [Result] Dishler JG, Slade S, Seifert S, Schallhorn SC. Small-Incision Lenticule Extraction (SMILE) for the Correction of Myopia with Astigmatism: Outcomes of the United States Food and Drug Administration Premarket Approval Clinical Trial. Ophthalmology. 2020 Aug;127(8):1020-1034. doi: 10.1016/j.ophtha.2020.01.010. Epub 2020 Jan 15. PMID 32173114